CLINICAL TRIAL: NCT06128382
Title: A First-in-human Phase 1, Single Center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Immunogenicity of Three Dose Levels of the OVX033 Vaccine, After Intramuscular Administration in Healthy Subjects Aged 18-49 Years
Brief Title: First-in-human Study to Evaluate the Safety and Immunogenicity of Three Dose Levels of the OVX033 Coronavirus Vaccine Candidate in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osivax (Industry)
Collaborators: CIC 1417 Cochin Pasteur Hôpital Cochin Paris France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: OVX033-001
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Dose escalation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- OVX033 - 100µg dose level (Experimental): Recombinant sarbecovirus vaccine based on the nucleocapsid of SARS-CoV-2. One single administration intramuscularly of a 100µg (0.2mL) dose on Day 1.
  Interventions: Biological: OVX033
- OVX033 - 250µg dose level (Experimental): Recombinant sarbecovirus vaccine based on the nucleocapsid of SARS-CoV-2. One single administration intramuscularly of a 250µg (0.5mL) dose on Day 1.
  Interventions: Biological: OVX033
- OVX033 - 500µg dose level (Experimental): Recombinant sarbecovirus vaccine based on the nucleocapsid of SARS-CoV-2. One single administration intramuscularly of a 500µg (1.0mL) dose on Day 1.
  Interventions: Biological: OVX033
- Saline solution - 0.2mL (Placebo Comparator): Saline solution (NaCl 0.9%), B. Braun Ecoflac® Plus 50mL. One single administration intramuscularly of a 0.2mL dose on Day 1.
  Interventions: Biological: Saline solution
- Saline solution - 0.5mL (Placebo Comparator): Saline solution (NaCl 0.9%), B. Braun Ecoflac® Plus 50mL. One single administration intramuscularly of a 0.5mL dose on Day 1.
  Interventions: Biological: Saline solution
- Saline solution - 1.0mL (Placebo Comparator): Saline solution (NaCl 0.9%), B. Braun Ecoflac® Plus 50mL. One single administration intramuscularly of a 1.0mL dose on Day 1.
  Interventions: Biological: Saline solution

INTERVENTIONS:
Biological: OVX033 — One single administration intramuscularly on Day 1
  Arms: OVX033 - 100µg dose level; OVX033 - 250µg dose level; OVX033 - 500µg dose level
Biological: Saline solution — One single administration intramuscularly on Day 1
  Arms: Saline solution - 0.2mL; Saline solution - 0.5mL; Saline solution - 1.0mL

SUMMARY:
This first-in-human clinical trial is designed to evaluate the safety and immunogenicity of one administration of OVX033 coronavirus vaccine at different dose levels (100µg, 250µg and 500µg)

DETAILED DESCRIPTION:
This trial is a first-in-human phase 1, single center, randomized, double-blind, placebo-controlled study in 48 adult subjects to evaluate the safety and immunogenicity of OVX033 sarbecovirus vaccine at different dose levels (100µg, 250µg and 500µg).

One single dose of OVX033 vaccine or of Placebo will be administered intramuscularly in healthy subjects aged 18-49 years.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Healthy male or female subjects, as determined by medical history and medical examination.
3. Aged 18 to 49 years.
4. Subjects who have been vaccinated (2 to 4 doses) with a licensed SARS-CoV-2 (COVID-19) vaccine. The last dose should be >6 months before administration of the investigational vaccine.
5. Reliable and willing to make themselves available for the duration of the study, willing and able to follow study procedures.
6. Willing to refrain from strenuous physical exercise during the week preceding any blood sampling, including between screening and vaccination visit (Visit 2).

Exclusion Criteria:

1. Subjects with a body mass index (BMI) <18 kg/m² or >30 kg/m² at screening.
2. Subjects weighing less than 50 kg.
3. Subjects with abnormal safety laboratory (hematology, biochemistry, coagulation and urinalysis) parameter at screening.
4. Subjects having previously received a non-licensed SARSCoV-2 vaccine or only one single dose of a licensed SARSCoV-2 vaccine.
5. Subjects having presented medically significant adverse event after having received a SARS-CoV-2 licensed vaccine.
6. Subjects currently treated with medications intended to prevent SARS-CoV-2 infection or disease (COVID-19) complications.
7. SARS-CoV-2 infection within the past 3 months prior to enrolment, RT-PCR-confirmed SARS-CoV-2 infection at screening or ongoing symptom of COVID-19.
8. Subjects having received another vaccination within 3 months prior to the day of study vaccination for live attenuated vaccines, or within 1 month prior to the day of study vaccination for inactivated vaccines.
9. Planning to receive other vaccines during the first 28 days following the study vaccine administration.
10. Female subjects: pregnant, breast-feeding or of childbearing potential without appropriate contraceptive methods in place for at least 2 months before enrolment, or with positive pregnancy test at screening or on the day of vaccination. Appropriate contraceptive methods are to be maintained until the end of the trial.
11. Subjects receiving treatment that can affect immune response such as systemic or high dose inhaled corticosteroids (>800μg/day beclomethasone or equivalent; occasional inhaled corticosteroids for asthma therapy are allowed), radiation treatment, cytotoxic drugs, or current or recent (within 3 months before study entry) chronic or prolonged (>10 days) use of systemic non-steroidal anti-inflammatory drugs, interferon, immunomodulators, allergy shots, as judged by the Investigator.
12. Any known or suspected immunodeficient conditions.
13. Past or current history of significant autoimmune diseases, as judged by the Investigator.
14. Known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) at screening.
15. Current history of medical illness such as diabetes, hypertension, heart, renal or hepatic diseases, as judged by the Investigator.
16. Hereditary or acquired hemorrhagic tendency or coagulation dysfunction (e.g., cytokine defects, coagulation disorders or platelet disorder), or history of serious bleeding, or history of massive bleeding after intramuscular injection, intravenous puncture or ecchymosis.
17. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of vaccination, or planned to receive such product during the whole study period.
18. Presence of an acute febrile illness on the day of planned vaccination or within 72 hours prior of it (oral temperature>38.0°C; temporary exclusion criterion).
19. Past or current history of any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
20. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
21. Past (stopped less than 6 months before enrolment) or current smoking habit above 10 cigarettes per day.
22. Past (stopped less than 6 months before enrolment) or current history of alcohol consumption (more than 2 glasses per day, more than 10 glasses per week, or absence of any days within a week without consumption. A standard glass contains 10 g of alcohol corresponding to 10 cl of wine, 25 cl of beer at 5% or 3 cl of alcohol at 40% [Société Française d'Alcoologie, 2023]).
23. Past (stopped less than 6 months before enrolment) or current history of use of recreational drugs.
24. Prophylactic or therapeutic use of any anti(retro)virals by systemic route during the study. Topical application is allowed.
25. History of severe allergic reactions and/or anaphylaxis, or serious adverse reactions to vaccines or allergy to kanamycin.
26. Any contraindication to intramuscular administration, as judged by the Investigator.
27. Individuals with history of any illness that, in the opinion of the Investigator, might interfere with the results of the study, or pose additional risk to the subjects due to participation in the study, either directly or through any treatments administered for that illness.
28. Sponsor employees or Investigator site personnel directly affiliated with this study, and their immediate families. Immediate family is defined as a spouse (or assimilated), parent, child or sibling, whether biological or legally adopted.
29. Subjects receiving ≥10 mg/day of prednisone or equivalent for more than 3 months before study entry.
30. Health professionals and/or students for whom vaccination against SARS-CoV-2 is strongly recommended.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Number and percentage of subjects reporting solicited local (Injection site redness, Injection site swelling, Injection site pain) and systemic (Fatigue, Headache, Arthralgia, Malaise, Myalgia, Fever) signs and symptoms | during 7 days after vaccine administration
Number and percentage of subjects reporting unsolicited adverse events | during 29 days after vaccine administration
Occurrence of adverse event of special interest | during the whole study duration, 180 days
Occurrence of serious adverse event | during the whole study duration, 180 days
Number and percentage of subjects with medically-attended adverse events (classified by type and reason) | during the whole study duration, 180 days
Number and percentage of subjects with deviations from normal values (judged clinically relevant or not by the Investigator) of safety laboratory tests | during 29 days after vaccine administration

SECONDARY OUTCOMES:
Cell-mediated immune response in terms of change of N-specific T-cell number in PBMCs, measured by IFNγ ELISPOT (after in vitro stimulation) | at Days 8, 29, 90 and 180 versus pre-injection baseline (Day 1)
N-specific CD4+ and CD8+T-cell percentages measured by flow cytometry (on PBMCs), identified as expressing markers (after in vitro stimulation), such as IL-2, TNFα and/or IFNγ | at Day 1 (pre-injection baseline) and Days 8 and 29
Geometric mean titers (GMTs) of anti-N IgG (ELISA, serum) | at Day 1 (pre-injection baseline), and Days 8, 29, 90 and 180
Number and percentage of subjects with an increase (four-fold) in anti-N IgG titer | on Days 8, 29, 90 and 180, with respect to preinjection baseline (Day 1)
Anti-OVX313 IgG (ELISA, serum) titers | at Days 29, 90 and 180 versus pre-injection baseline (Day 1)
anti-hC4BP oligomerization domain IgG (ELISA, serum) titers [If positive result for anti-OVX313] | at Days 29, 90 and 180 versus pre-injection baseline (Day 1)
Number and percentage of subjects with a RT-PCR-confirmed SARS-CoV-2 and/or influenza A or B infection | during the whole study duration, 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Odile Launay, MD, Principal Investigator — CIC Cochin Pasteur CIC 1417 Hôpital Cochin
Locations (1):
- CIC Cochin Pasteur CIC 1417 Hôpital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No